CLINICAL TRIAL: NCT06772922
Title: Effects of a Pulmonary and Cardiovascular Rehabilitation Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Letícia Baltieri, Physiotherapist at CECOM-UNICAMP, PhD in Sciences, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4.004.580
Record Dates: First submitted 2025-01-07; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Muscle Weakness; Quality of Lifte; Dyspnea; Asthmatic; Dyspnea; Cardiac; Dyspnea
Keywords: pulmonary rehabilitation; Non-communicable chronic diseases; cardiovascular disease; cardiac rehabilitation
MeSH Terms: conditions — Dyspnea; Asthma; Noncommunicable Diseases; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise (Other)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — effect of exercise after three months (comparison of the patient with himself)

SUMMARY:
Non-communicable chronic diseases (NCDs) affect approximately 30% of the adult global population, significantly impacting respiratory function and quality of life. Pulmonary and cardiovascular rehabilitation has proven to be an effective therapeutic intervention for managing respiratory symptoms and cardiovascular and improving functional capacity in patients with chronic respiratory conditions. The objective of this study is to evaluate the effects of the pulmonary and cardiovascular rehabilitation program on users of the physical therapy service of CECOM of UNICAMP related to functional capacity, quality of life and respiratory variables after 3 months of the program. Candidates for the pulmonary rehabilitation program are users diagnosed with chronic obstructive pulmonary disease (COPD), pulmonary emphysema, pulmonary fibrosis, asthma or other lung disease. Candidates for the cardiovascular rehabilitation program are users diagnosed with: infarction (AMI), myocardial revascularization surgery, coronary angioplasty, stable angina, valve replacement, chronic heart failure and who meet the criteria for phase III of cardiovascular rehabilitation. They should be referred to physical therapy by the cardiologist with complementary exams and exercise test. The program's assessment will consist of: anamnesis, analysis and recording of complementary exams, physical assessment (weight, height, BMI, cardiac and pulmonary auscultation, blood pressure, heart rate, peripheral oxygen saturation, respiratory muscle strength), functional capacity (six-minute walk test) and quality of life (questionnaire). The program will include aerobic exercises on a treadmill or stationary bike with an intensity between 50-70% of the reserve HR, below the ischemic thresholds. It will also include peripheral muscle strength exercises for the upper and lower limbs, in addition to respiratory muscle training for lung disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for the pulmonary rehabilitation program: users diagnosed with chronic obstructive pulmonary disease (COPD), pulmonary emphysema, pulmonary fibrosis, asthma or other lung disease.
* Candidates for the cardiovascular rehabilitation program: users diagnosed with acute myocardial infarction, myocardial revascularization surgery, coronary angioplasty, stable angina, valve replacement, chronic heart failure and who meet the criteria for phase III of cardiovascular rehabilitation.
* Referral with medical clearance for rehabilitation

Exclusion Criteria:

* Patients with any contraindication to aerobic or muscle-strengthening physical exercise, such as significant arrhythmias, untreated heart disease, myocarditis, recent or untreated pulmonary embolism, and uncontrolled systemic arterial hypertension, among other conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-03-03 (Actual); Primary Completion 2024-11-03 (Actual); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Functional Capacity | three months
  The Six-Minute Walk Test (6MWT) is used to measure functional capacity. For the test, the study participant walks in a flat 30-meter corridor for 6 minutes and the evaluator marks the final distance covered. This distance is normalized according to age and individual anthropometric characteristics in a solution validated in the literature. This distance represents the functional capacity that can be within or below that predicted by the literature.
Inspiratory muscle strength | three months
  Using an analog manometer, inspiratory muscle strength was assessed by means of maximum inspiratory pressure (MIP) in cmH2O. During this procedure, the patient was comfortably seated in a chair with his/her feet flat on the floor and, using a nose clip, was instructed to take a maximal deep inspiration into the mouthpiece of the device after a complete exhalation. The average of three dimensions was recorded. Both the absolute value of the estimates and the predicted value according to the literature were recorded using the following equations according to Neder et al., 1999
Expiratory muscle strength | three months
  Using an analog manometer, exspiratory muscle strength was assessed by means of maximum inspiratory pressure (MEP) in cmH2O. During this procedure, the patient was comfortably seated in a chair with his/her feet flat on the floor and, using a nose clip, was instructed to take a maximal deep expiration into the mouthpiece of the device after a complete inspiration. The average of three dimensions was recorded. Both the absolute value of the estimates and the predicted value according to the literature were recorded using the following equations according to Neder et al., 1999

SECONDARY OUTCOMES:
Quality of life | three months
  We will use the St. George's Respiratory Questionnaire or SF-36

CONTACTS AND LOCATIONS:
Locations (1):
- Unicamp, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No